CLINICAL TRIAL: NCT06811129
Title: Long-Term Neurologic and Neurocognitive Sequelae Following Pediatric Ebola Virus in Liberia
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001809; 001809-N
Record Dates: First submitted 2025-02-05; First posted 2025-02-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-02-10

CONDITIONS: Ebola; Post-Acute Ebola Syndrome
Keywords: Ebola; Neurologic; Pediatric; Post-Acute Ebola Syndrome; Cognitive; Global Neurology
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Close Contacts: Male of female, previously enrolled in PREVAIL III Natural History of Ebola study as a close contact. Close contacts are those who had a relationship with someone who survived EVD but were never diagnosed with EVD themselves.
- EVD Survivors: Male or female, previously enrolled in PREVAIL III Natural History of Ebola study as an EVD survivor.

SUMMARY:
Background:

Ebola virus disease (EVD) causes fever, vomiting, and diarrhea, and may cause internal bleeding. It is often fatal. EVD may also damage the brain and nervous system. It can cause headaches, tremors, weakness, and other problems. These issues can continue for years after people recover from EVD infection. Researchers want to understand more about how EVD may have affected the brains of people who contracted the disease as children.

Objective:

To learn more about the long-term effects of EVD on the brain and nervous system in people who had the disease as children.

Eligibility:

People who were less than 18 years old when they took part in a previous study called the PREVAIL III Natural History of Ebola study. They can be either a survivor of EVD or a close contact. A close contact is someone who had a relationship with a person who survived EVD but never had the disease themself.

Design:

Participants will have 1 clinic visit. They will undergo several tasks:

They will have an exam of their nervous system performed by a neurologist. They will do physical tasks and answer questions about any problems or symptoms since they had EVD.

They may have blood drawn.

They will have tests of their memory, attention, and thinking skills. For one test, participants will answer questions and solve puzzles using pencil and paper. For another test, they will play 4 different games on an iPad.

They will have an interview. A researcher will ask questions about their mood and other symptoms that may affect their brain and nervous system; their past medical diagnoses, symptoms, and experiences; and how they are doing at home, school, or work.

DETAILED DESCRIPTION:
Study Description:

The long-term neurological sequelae of Ebola virus disease (EVD) are not well-described, particularly in survivors infected during pediatric age. The 2015 west Africa EVD epidemic had dramatic effect on adults and children and by one year following infection, concerns for neurologic sequelae became apparent. The PREVAIL III (PIII) Ebola Natural History Study in Monrovia, Liberia had a number of substudies, including both an adult Neurology and pediatric Neurology Substudy which were undertaken to better understand the long-term neurologic sequelae of EVD. The adult Neurology Substudy had over five years of follow up visits whereas the original Pediatric Neurology Substudy cohort was composed of a small sample of children seen in 2015 one time under PIII with no subsequent follow ups. Although this pediatric cohort was small, pilot data from this assessment revealed lower cognitive scores in the pediatric EVD survivors compared to controls, as well as worse executive function scores, more complaints of neuropsychiatric symptoms, and worse disability on modified Rankin Scale, among other findings. PIII subsequently closed out between 2020 and 2021. Here we propose a new protocol to observe and study the neurologic and neurocognitive sequelae following Ebola virus exposure at an age below 18. We propose conducting a single in-person neurologic visit including neurologic exam, neurocognitive assessment, and neurologic history and symptom questionnaire to be given to participants at greater than 5-years following exposure. We also plan to do a single blood draw at time of visit to assess for Ebola Virus antibody titers in survivors and close contacts (controls). The participants included in this study will include Ebola survivors and close contacts (controls) that were enrolled in PIII at age less than 18. We hypothesize that some pediatric Ebola survivors will have longterm neurologic sequelae at greater than 5 years post exposure that may be subtle in nature. Included in this study will be one embedded substudy.

Longitudinal Pediatric Neuro EVD Substudy: We propose to see the original small cohort of pediatric participants seen in 2015 for a second visit as a longitudinal sub study. In evaluating our longitudinal cohort, we expect that some of the sequelae noted during their initial evaluation may have improved over time, but these survivors still may have persistent neurological sequelae even after over 5 years convalescence from EVD.

Objectives:

Primary Objective:

1. Pediatric EVD Neuro Follow up Study: To observe and describe the range of neurologic and neurocognitive findings that are present in EVD survivors at greater than 5 years following infection as compared to controls.
2. Longitudinal Pediatric Neuro EVD Substudy (Subset of population): To compare neurologic and neurocognitive findings found in EVD survivors and controls at greater than 5 years following infection to that of the same participants at first visit about 1 year post infection.

Secondary Objectives

1. Pediatric EVD Neuro Follow up Study: To characterize serum Zaire Ebola virus (EBOV) specific antibodies in pediatric EVD survivors at greater than 5 years following infection compared to that of controls.
2. Longitudinal Pediatric Neuro EVD Substudy: To characterize serum EBOV specific antibodies in pediatric EVD survivors at greater than 5 years following infection to that of the same participant at first visit about 1 year post infection.

Exploratory Objective:

Pediatric EVD Neuro Follow up Study

1. To compare EBOV specific antibodies in pediatric EVD survivors with and without neurologic and neurocognitive sequelae.
2. To compare neurologic and neurocognitive findings in pediatric EVD survivors and controls at greater than 5 years post infection to that of adult participants from the PIII adult Neurology sub study.
3. To explore the presence of other serologic markers in pediatric EVD survivors compared to close-contacts (control).

Outcomes:

Primary Endpoint:

1. Pediatric EVD Neuro Follow up Study: In comparison of EVD survivors at greater than 5 years following infection with close contacts (controls), the prevalence of:

   * neurological symptoms (as asked on neurologic symptom questionnaire CRF)
   * physical disability (as assessed through MRS score)
   * executive function dysfunction (as assessed through executive function assessment questions)
   * neuropsychiatric symptoms (as indicated on neuropsychiatric symptom portion of CRF)
   * neurologic exam abnormalities (as found on full neurologic physical exam performed by licensed neurologist during visit)
   * neurocognitive deficits (as determined by cognitive exam scores on NIH Toolbox exam and ICA-P assessment)
2. Longitudinal Pediatric Neuro EVD Substudy: In comparison of EVD survivors at greater than 5 years following infection to that at first visit about 1 year after infection, the change in:

   * number of neurological symptoms (as asked on neurologic symptom questionnaire CRF)
   * Physical disability (as assessed through MRS score)
   * Executive function dysfunction (as assessed through executive function assessment questions).
   * number of neuropsychiatric symptoms (as indicated on neuropsychiatric symptom portion of CRF.
   * persistence of neurologic exam abnormalities (as found on full neurologic physical exam performed by licensed neurologist during visit).
   * neurocognitive deficits (as determined by cognitive exam scores on NIH Toolbox exam and ICA-P assessment).

Secondary Endpoints:

1. Pediatric EVD Neuro Follow up Study: The degree of antibody response in pediatric EVD survivors at greater than 5 years following infection compared to that of close contacts (controls).
2. Longitudinal Pediatric Neuro EVD Substudy: The degree of antibody response in pediatric EVD survivors at greater than 5 years following infection compared to that at about 1 year following infection.

Exploratory Endpoints:

Pediatric EVD Neuro Follow up Study:

1. In EVD survivors at greater than 5 years post infection, the correlation between serum EBOV specific antibody presence and:

   * presence of neurological symptoms (as asked on neurologic symptom questionnaire CRF).
   * presence of physical disability (as assessed through MRS score).
   * presence of executive function dysfunction (as assessed through executive function assessment questions)
   * presence of neuropsychiatric symptoms (as indicated on neuropsychiatric symptom portion of CRF)
   * presence of neurologic exam abnormalities (as found on full neurologic physical exam performed by licensed neurologist during visit).
   * presence of neurocognitive deficits (as determined by cognitive exam scores on NIH Toolbox exam)
2. In pediatric versus adult EVD survivors at greater than 5 years following infection, the prevalence of:

   * neurological symptoms (as asked on neurologic symptom questionnaire CRF).
   * physical disability (as assessed through MRS score)
   * neuropsychiatric symptoms (as indicated on neuropsychiatric symptom portion of CRF)
   * neurologic exam abnormalities (as found on full neurologic physical exam performed by licensed neurologist during visit)
   * neurocognitive deficits (as determined by cognitive exam scores on NIH Toolbox exam).
3. The profile of serologic immune markers in pediatric EVD survivors at greater than 5 years following infection.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Male or female, previously enrolled in PREVAIL III Natural History of Ebola study as either an EVD survivor, or a close contact.*
3. Aged < 18 Years Old at the time of enrollment in PREVAIL III Natural History of Ebola study.
4. Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

   * Close contacts are those who had a relationship with someone who survived EVD but were never diagnosed with EVD themselves.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. At the time of enrollment, lacks consent capacity due to cognitive impairment that would make them incapable of understanding the explanation of the procedures in this study. Cognitive capacity to consent will be determined at the time of enrollment. Participants with mental disorders or those participants who are cognitively impaired yet still retain consent capacity will not be excluded.
2. Is unable to comply with the procedures of the protocol.
3. Has any condition in the judgement of the study staff that would make the volunteer unable to participate in the study.
4. Is non-English speaking.

Justification for the Exclusion of Non-English Speakers

We plan to include speakers of simple Liberian English in this study. The tools we use for cognitive testing are not validated in any other language, other than English. It is expected that most, if not all, of the cohort we will be recruiting from will be simple Liberian English speakers.

Ages: 7 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will include participants of the PREVAIL III Natural History of Ebola Study who were of pediatric age at the time of enrollment, including EVD survivors and close contacts.
Sampling Method: Non-Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2026-01-29 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Pediatric EVD Neuro Follow up Study | 5-10 years post-infection
  To observe and describe the range of neurologic and neurocognitive findings that are present in EVD survivors at greater than 5 years following infection as compared to controls. In comparison of EVD survivors at greater than 5 years following infection with close contacts, the prevalence of:- neurological symptoms (as asked on neurologic symptom questionnaire CRF) - physical disability (as assessed through MRS score) - executive function dysfunction (as assessed through executive function assessment questions) - neuropsychiatric symptoms (as indicated on neuropsychiatric symptom portion of CRF) - neurologic exam abnormalities (as found on full neurologic physical exam performed by licensed neurologist during visit) - neurocognitive deficits (as determined by cognitive exam scores on NIH Toolbox exam and ICA-P assessment)
Longitudinal Pediatric Neuro EVD Sub study (Subset of population) | 5-10 years post-infection
  To compare neurologic and neurocognitive findings found in EVD survivors and controls at greater than 5 years following infection to that of the same participants at first visit about 1 year post infection.- number of neurological symptoms (as asked on neurologic symptom questionnaire CRF) - Physical disability (as assessed through MRS score) - Executive function dysfunction (as assessed through executive function assessment questions).- number of neuropsychiatric symptoms (as indicated on neuropsychiatric symptom portion of CRF.- persistence of neurologic exam abnormalities (as found on full neurologic physical exam performed by licensed neurologist during visit).- neurocognitive deficits (as determined by cognitive exam scores on NIH Toolbox exam and ICA-P assessment).

SECONDARY OUTCOMES:
Longitudinal Pediatric Neuro EVD Sub study: | 5-10 years post-infection
  The degree of antibody response in pediatric EVD survivors after 5 years or more of convalescence from EVD compared to that at 1 year following infection.
Pediatric EVD Neuro Follow up Study | 5-10 years post-infection
  The degree of antibody response in pediatric EVD survivors after 5 years or more of convalescence from EVD compared to that of controls.

CONTACTS AND LOCATIONS:
Overall Officials: Bridgette J Billioux, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- John F. Kennedy Medical Center, Monrovia, Liberia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bwaka MA, Bonnet MJ, Calain P, Colebunders R, De Roo A, Guimard Y, Katwiki KR, Kibadi K, Kipasa MA, Kuvula KJ, Mapanda BB, Massamba M, Mupapa KD, Muyembe-Tamfum JJ, Ndaberey E, Peters CJ, Rollin PE, Van den Enden E, Van den Enden E. Ebola hemorrhagic fever in Kikwit, Democratic Republic of the Congo: clinical observations in 103 patients. J Infect Dis. 1999 Feb;179 Suppl 1:S1-7. doi: 10.1086/514308. PMID 9988155
- [Background] Clark DV, Kibuuka H, Millard M, Wakabi S, Lukwago L, Taylor A, Eller MA, Eller LA, Michael NL, Honko AN, Olinger GG Jr, Schoepp RJ, Hepburn MJ, Hensley LE, Robb ML. Long-term sequelae after Ebola virus disease in Bundibugyo, Uganda: a retrospective cohort study. Lancet Infect Dis. 2015 Aug;15(8):905-12. doi: 10.1016/S1473-3099(15)70152-0. Epub 2015 Apr 21. PMID 25910637
- [Background] Schieffelin JS, Shaffer JG, Goba A, Gbakie M, Gire SK, Colubri A, Sealfon RS, Kanneh L, Moigboi A, Momoh M, Fullah M, Moses LM, Brown BL, Andersen KG, Winnicki S, Schaffner SF, Park DJ, Yozwiak NL, Jiang PP, Kargbo D, Jalloh S, Fonnie M, Sinnah V, French I, Kovoma A, Kamara FK, Tucker V, Konuwa E, Sellu J, Mustapha I, Foday M, Yillah M, Kanneh F, Saffa S, Massally JL, Boisen ML, Branco LM, Vandi MA, Grant DS, Happi C, Gevao SM, Fletcher TE, Fowler RA, Bausch DG, Sabeti PC, Khan SH, Garry RF; KGH Lassa Fever Program; Viral Hemorrhagic Fever Consortium; WHO Clinical Response Team. Clinical illness and outcomes in patients with Ebola in Sierra Leone. N Engl J Med. 2014 Nov 27;371(22):2092-100. doi: 10.1056/NEJMoa1411680. Epub 2014 Oct 29. PMID 25353969
- [Background] Chertow DS, Nath A, Suffredini AF, Danner RL, Reich DS, Bishop RJ, Childs RW, Arai AE, Palmore TN, Lane HC, Fauci AS, Davey RT. Severe Meningoencephalitis in a Case of Ebola Virus Disease: A Case Report. Ann Intern Med. 2016 Aug 16;165(4):301-4. doi: 10.7326/M15-3066. Epub 2016 Apr 5. No abstract available. PMID 27043004
- [Background] Howlett P, Brown C, Helderman T, Brooks T, Lisk D, Deen G, Solbrig M, Lado M. Ebola Virus Disease Complicated by Late-Onset Encephalitis and Polyarthritis, Sierra Leone. Emerg Infect Dis. 2016 Jan;22(1):150-2. doi: 10.3201/eid2201.151212. No abstract available. PMID 26690042
- [Background] Jacobs M, Rodger A, Bell DJ, Bhagani S, Cropley I, Filipe A, Gifford RJ, Hopkins S, Hughes J, Jabeen F, Johannessen I, Karageorgopoulos D, Lackenby A, Lester R, Liu RS, MacConnachie A, Mahungu T, Martin D, Marshall N, Mepham S, Orton R, Palmarini M, Patel M, Perry C, Peters SE, Porter D, Ritchie D, Ritchie ND, Seaton RA, Sreenu VB, Templeton K, Warren S, Wilkie GS, Zambon M, Gopal R, Thomson EC. Late Ebola virus relapse causing meningoencephalitis: a case report. Lancet. 2016 Jul 30;388(10043):498-503. doi: 10.1016/S0140-6736(16)30386-5. Epub 2016 May 18. PMID 27209148
- [Background] Fallah MP, Reilly C, Van Ryn C, Badio M, Camanor SW, Kaler SG, Johnson B, Orone R, Flumo H, Moses SJ, Johnson KL, Gorpudolo N, Gayedyu-Dennis D, Dighero-Kemp B, Fayiah J, Marron L, Hensley LE, Taylor RJ, Higgs ES, Lane HC, Neaton JD, Sneller MC. Pregnancy, pregnancy outcomes, and infant growth and development after recovery from Ebola virus disease in Liberia: an observational cohort study. Lancet Glob Health. 2023 Jul;11(7):e1053-e1060. doi: 10.1016/S2214-109X(23)00210-3. PMID 37349033
- [Background] Foeller ME, Carvalho Ribeiro do Valle C, Foeller TM, Oladapo OT, Roos E, Thorson AE. Pregnancy and breastfeeding in the context of Ebola: a systematic review. Lancet Infect Dis. 2020 Jul;20(7):e149-e158. doi: 10.1016/S1473-3099(20)30194-8. Epub 2020 May 6. PMID 32595045
- [Background] PREVAIL III Study Group; Sneller MC, Reilly C, Badio M, Bishop RJ, Eghrari AO, Moses SJ, Johnson KL, Gayedyu-Dennis D, Hensley LE, Higgs ES, Nath A, Tuznik K, Varughese J, Jensen KS, Dighero-Kemp B, Neaton JD, Lane HC, Fallah MP. A Longitudinal Study of Ebola Sequelae in Liberia. N Engl J Med. 2019 Mar 7;380(10):924-934. doi: 10.1056/NEJMoa1805435. PMID 30855742
- [Background] Diallo MSK, Ayouba A, Keita AK, Thaurignac G, Sow MS, Kpamou C, Barry TA, Msellati P, Etard JF, Peeters M, Ecochard R, Delaporte E, Toure A; PostEbogui Study Group. Temporal evolution of the humoral antibody response after Ebola virus disease in Guinea: a 60-month observational prospective cohort study. Lancet Microbe. 2021 Dec;2(12):e676-e684. doi: 10.1016/S2666-5247(21)00170-1. Epub 2021 Sep 3. PMID 35544108